CLINICAL TRIAL: NCT04319094
Title: Peer Enhanced Depression Care: Using Peer Mentors to Provide Self Care Support to Low Income and Minority Older Adults
Brief Title: PEERS Using Peer Mentors to Deliver Depression Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jin hui Joo, MD, MA, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022P001675; R01MH123165 (NIH)
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEERS (Experimental): Peer mentors who have experience of depression are trained and supervised to deliver depression care. Peers will meet with depressed older adults for 8 weekly meeting lasting approximately 45 minutes. Peer mentors will provide social support defined as emotional, informational and appraisal support that includes coping strategies. Peers will be supervised by a mental health professional.
  Interventions: Behavioral: PEERS
- Social interaction (Active Comparator): A study staff member will provide eight weekly social interaction visits and phone calls to the depressed older adult.
  Interventions: Other: Social interaction

INTERVENTIONS:
Behavioral: PEERS — Peer mentors deliver depression care that include social support and coping skills, focused on goal setting and small behavioral changes.
  Arms: PEERS
Other: Social interaction — Study staff will provide a combination of 8 social interaction visits and phone calls to the participants randomized to this condition.
  Arms: Social interaction

SUMMARY:
Fifteen to twenty percent of older Americans (6 to 8 million people) suffer from depression but more than one-half do not receive any services, a burden disproportionately shared by low-income and minority older adults who receive few or no services. The investigators propose to test a community-based peer model of depression care called PEERS (a peer support program) that provides self-care support for minority and low-income older adults.

DETAILED DESCRIPTION:
Depression is a major burden for minority and low-income older adults who are less likely to use mental health services, and development of new service delivery models is needed to improve the quality of life and address disparities to access for this group. The investigators propose to test the effectiveness of a peer-delivered depression care program that is embedded in the community and linked to the patient's primary care clinic. The investigators will carry out a randomized controlled trial of the PEERS program in which peer mentors who have personal experience of depression meet individually with older adults recruited in the community for 8 weekly meetings focused on relief of depressive symptoms through self-care support and linkages to community resources. This group of low-income and minority older adults in the intervention will be compared to a group that receives non-peer visits that provide social interaction. The PEERS program takes a chronic disease self-management approach and is guided by the conceptual frameworks of social support, peer support, and social learning. The investigators will conduct an analysis of mediation to understand the mechanism of peer support, by measuring factors such as self-efficacy and loneliness that may be responsible for the intervention effect. The investigators' goal is to use peer-delivered depression care to decrease the mental health morbidity of at-risk low-income and minority adults. The potential public health impact is high because the investigators' project seeks to increase access to depression for a vulnerable group of older adults who often do not get care and leverages an existing workforce of peer workers whose services are reimbursed in many states.

ELIGIBILITY:
Inclusion Criteria:

* 50 years and older
* depressive symptoms with Patient Health Questionnaire-9 scores ≥ 5
* belong to an underserved population, defined as annual income less than 200% of the federal poverty level ($24,120) and/or self-identified ethnic minority
* able to communicate in English
* willing to give informed consent.

Exclusion Criteria:

* meet diagnostic criteria for mania or hypomania
* meet diagnostic criteria for psychotic syndrome
* meet diagnostic criteria for substance abuse or dependence
* acutely suicidal
* a score on the Mini-Mental State Examination (MMSE) ≤ 24
* currently taking an antidepressant medication with dosage change in the past 3 months
* receiving active psychotherapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Joo JH, Xie A, Choi N, Gallo JJ, Zhong Y, Ma M, Locascio JJ, Khemraj U, Mace RA, Solomon P. A Mixed Methods Effectiveness Study of a Peer Support Intervention for Older Adults During the COVID-19 Pandemic: Results of a Randomized Clinical Trial. Am J Geriatr Psychiatry. 2025 Apr;33(4):389-401. doi: 10.1016/j.jagp.2024.09.013. Epub 2024 Oct 10. PMID 39438236

RESULTS

PARTICIPANT FLOW:
Groups:
- PEERS: Peer mentors who have experience of depression are trained and supervised to deliver depression care. Peers will meet with depressed older adults for 8 weekly meeting lasting approximately 45 -60 minutes. Peer mentors will provide social support defined as emotional, informational and appraisal support that includes coping strategies. Peers will be supervised by a mental health professional.
  PEERS: Peer mentors deliver depression care that include social support and coping skills, focused on goal setting and small behavioral changes.
- Social Interaction: A study staff member will provide eight weekly social interaction phone calls to the depressed older adult.
  Social interaction: Study staff will provide a social interaction phone calls to the participants randomized to this condition.
Period: Baseline
Arm/Group | PEERS | Social Interaction
Started | 75 | 74
Completed | 69 | 65
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 4 | 5
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1
Period: Post-Intervention
Arm/Group | PEERS | Social Interaction
Started | 69 | 65
Completed | 56 | 52
Not Completed | 13 | 13
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Incomplete Data Collection | 1 | 3
Period: 3-month
Arm/Group | PEERS | Social Interaction
Started | 57 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.) | 55 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.)
Completed | 45 | 43
Not Completed | 12 | 12
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Incomplete data collection | 9 | 7
Period: 6-month
Arm/Group | PEERS | Social Interaction
Started | 54 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.) | 50 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.)
Completed | 39 | 37
Not Completed | 15 | 13
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Incomplete data collection | 14 | 9
Period: 9-month
Arm/Group | PEERS | Social Interaction
Started | 53 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.) | 46 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.)
Completed | 37 | 36
Not Completed | 16 | 10
Not completed — Lost to Follow-up | 8 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Incomplete data collection | 8 | 5
Period: 12-month
Arm/Group | PEERS | Social Interaction
Started | 45 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.) | 41 (Participants who did not complete data collection for a previous period can continue and provide data in the next period.)
Completed | 34 | 33
Not Completed | 11 | 8
Not completed — Lost to Follow-up | 11 | 8

BASELINE CHARACTERISTICS:
Population: Baseline analysis population consists of participants randomized to one of the study arm and completed baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PEERS | Social Interaction | Total
Number analyzed (Participants) | 69 | 65 | 134
Age, Continuous [Median (Full Range); unit: Years] | 69.0 [54.0 to 95.0] | 70.0 [51.0 to 94.0] | 69.5 [51.0 to 95.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 113
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 66 | 65 | 131
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 35 | 70
  White | 27 | 28 | 55
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 69 | 65 | 134
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — Depression will be assessed with the Patient Health Questionnaire (PHQ)-9. The PHQ-9 score is summed. There are 9 items in the questionnaire and scores range from 0 to 27. A score of 5 indicates mild depressive symptoms, 10 - 14 indicates moderate depression, 15-19 indicates moderately severe depression, 20-27 indicates severe depression.
  units on a scale | 10.81 (4.88) | 10.4 (4.7) | 10.6 (4.78)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-9
Description: Depression will be assessed with the Patient Health Questionnaire (PHQ)-9. The PHQ-9 score is summed. There are 9 items in the questionnaire and scores range from 0 to 27. A score of 5 indicates mild depressive symptoms, 10 - 14 indicates moderate depression, 15-19 indicates moderately severe depression, 20-27 indicates severe depression.
Time Frame: Baseline, post-intervention (8-week), 3 months after intervention, 6 months after intervention, 9 months after intervention, 12 months after intervention
Population: All participants with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
score on a scale
  Post-intervention: number analyzed (Participants) | 56 | 52
  Post-intervention | 6.66 (4.51) | 7.33 (4.28)
  3 Months: number analyzed (Participants) | 45 | 43
  3 Months | 7.89 (4.91) | 7.84 (4.73)
  6 Months: number analyzed (Participants) | 38 | 37
  6 Months | 7.95 (4.81) | 8.03 (5.35)
  9 Months: number analyzed (Participants) | 39 | 36
  9 Months | 8.77 (5.57) | 7.14 (4.57)
  12 Months: number analyzed (Participants) | 33 | 33
  12 Months | 8.09 (5.05) | 8.42 (5.01)
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores from baseline to post-intervention for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 501; Mean Difference (Net) = -3.7, 95% CI 2-sided [-4.77 to -2.62], Standard Error of Mean 0.55 — Score difference = Post-intervention - Baseline; A series of generalized linear mixed-effect models were implemented to predict the outcome measurements. The primary fixed effect predictors were group (control vs. PEERS), time (categorical), and group * time. Random terms in all models were: study participants and their interaction with time. The covariance of dependent variable values across time was modeled as a first-order auto-regression decaying function (AR1). Higher order fixed and random terms were pretested and removed from the model if nonsignificant
Statistical Analysis 2: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores from baseline to 3-month for all study participants; Test type: Superiority; p = 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 501; Mean Difference (Net) = -2.53, 95% CI 2-sided [-3.81 to -1.25], Standard Error of Mean 0.65 — Score difference = 3-month - Baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores from baseline to 6-month for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 501; Median Difference (Net) = -2.83, 95% CI 2-sided [-4.13 to -1.53], Standard Error of Mean 0.66 — Score difference = 6-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores from baseline to 9-month for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 501; Mean Difference (Net) = -2.76, 95% CI 2-sided [-4.03 to -1.49], Standard Error of Mean 0.65 — Score difference = 9-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Patient Health Questionnaire-9 (PHQ-9) scores from baseline to 12-month for all study participants; Test type: Superiority; p = 0.0003, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 501; Mean Difference (Net) = -2.56, 95% CI 2-sided [-3.95 to -1.17], Standard Error of Mean 0.71 — Score difference =12-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: PEERS vs Social Interaction; Null hypothesis: There is no difference in the change of PHQ-9 over time between the control and PEERS participants; Test type: Superiority; p = 0.4375, Mixed Models Analysis

2. Secondary Outcome: Rand Health Survey Short Form 36 - Physical Functioning
Description: The RAND 36-Item Health Survey is a set of generic, coherent, and easily administered quality-of-life measures. Each item is scored on a 0 to 100 range. Higher scores indicate better functioning.The physical functioning subscale was calculated using the average of 10 of the 36 items (item 3, 4, 5, 6, 7, 8, 9, 10, 11, 12)
Time Frame: Baseline, post-intervention (8-week), 3 months after intervention , 6 months after intervention, 9 months after intervention, 12 months intervention
Population: All participants with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
score on a scale
  Post-Intervention: number analyzed (Participants) | 53 | 51
  Post-Intervention | 47.64 (28.82) | 50 (30.07)
  3 Month: number analyzed (Participants) | 42 | 40
  3 Month | 50.12 (29.02) | 50.88 (30.57)
  6 Month: number analyzed (Participants) | 33 | 32
  6 Month | 43.48 (27.34) | 49.69 (29.13)
  9 Month: number analyzed (Participants) | 33 | 33
  9 Month | 46.06 (30.36) | 50.3 (30.72)
  12 Month: number analyzed (Participants) | 26 | 28
  12 Month | 49.62 (26.09) | 44.46 (29.04)
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36 - Physical Functioning scores from baseline to post-intervention for all study participants; Test type: Superiority; p = 0.51, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 364; Mean Difference (Net) = 1.61, 95% CI 2-sided [-3.15 to 6.37], Standard Error of Mean 2.42; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-physical function scores from baseline to 3-month for all study participants; Test type: Superiority; p = 0.18, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 364; Mean Difference (Net) = 4.57, 95% CI 2-sided [-2.08 to 11.21]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-physical function scores from baseline to 6-month for all study participants; Test type: Superiority; p = 0.63, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 364; Mean Difference (Net) = 1.57, 95% CI 2-sided [-4.89 to 8.04], Standard Error of Mean 3.29; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-physical function scores from baseline to 9-month for all study participants; Test type: Superiority; p = 0.74, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 364; Mean Difference (Net) = -1.02, 95% CI 2-sided [-6.94 to 4.91], Standard Error of Mean 3.01; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-physical function scores from baseline to 12-month for all study participants; Test type: Superiority; p = 0.85, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 364; Mean Difference (Net) = 0.7, 95% CI 2-sided [-6.82 to 8.23], Standard Error of Mean 3.83; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: PEERS vs Social Interaction; Null hypothesis: There is no difference in the change of physical functioning over time between the control and PEERS participants; Test type: Superiority; p = 0.3988, Mixed Models Analysis

3. Secondary Outcome: Rand Health Survey Short Form 36 Item - Social Functioning
Description: The RAND 36-Item Health Survey is a set of generic, coherent, and easily administered quality-of-life measures. Each item is scored on a 0 to 100 range. Higher scores indicate better functioning. The social functioning subscale was calculated using the average of 2 of the 36 items (item 20, 32)
Time Frame: as for outcome 2
Population: All participants with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
score on a scale
  Post-intervention: number analyzed (Participants) | 51 | 51
  Post-intervention | 60.29 (30.18) | 59.56 (25.32)
  3 Month: number analyzed (Participants) | 42 | 40
  3 Month | 64.29 (32.26) | 66.88 (26.18)
  6 Month: number analyzed (Participants) | 33 | 31
  6 Month | 59.47 (25.59) | 63.71 (28.75)
  9 Month: number analyzed (Participants) | 32 | 33
  9 Month | 38.75 (28.58) | 60.61 (32.79)
  12 Month: number analyzed (Participants) | 26 | 29
  12 Month | 5.73 (61.54) | 53.88 (28.76)
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-social function scores from baseline to post-intervention for all study participants; Test type: Superiority; p = 0.14, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 360; Mean Difference (Net) = 5.08, 95% CI 2-sided [-1.63 to 11.79], Standard Error of Mean 3.41; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-social function scores from baseline to 3-month for all study participants; Test type: Superiority; p = 0.01, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 360; Mean Difference (Net) = 10.32, 95% CI 2-sided [2.45 to 18.19], Standard Error of Mean 4; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-social function scores from baseline to 6-month for all study participants; Test type: Superiority; p = 0.015, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 360; Mean Difference (Net) = 10.25, 95% CI 2-sided [2.01 to 18.5], Standard Error of Mean 4.19; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-social function scores from baseline to 9-month for all study participants; Test type: Superiority; p = 0.004, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; degrees of freedom: 360; Mean Difference (Net) = 11.72, 95% CI 2-sided [3.7 to 19.73], Standard Error of Mean 4.07; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-social function scores from baseline to 12-month for all study participants; Test type: Superiority; p = 0.2, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 360; Mean Difference (Net) = 5.73, 95% CI 2-sided [-3.09 to 14.55], Standard Error of Mean 4.49; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: PEERS vs Social Interaction; Null hypothesis: There is no difference in the change of social functioning over time between the control and PEERS participants; Test type: Superiority; p = 0.8037, Mixed Models Analysis

4. Secondary Outcome: Rand Health Survey Short Form 36 Item - Emotional Functioning
Description: The RAND 36-Item Health Survey is a set of generic, coherent, and easily administered quality-of-life measures. Each item is scored on a 0 to 100 range. Higher scores indicate better functioning. The emotional functioning subscale was calculated using the average of 3 of the 36 items (item 17, 18, 19)
Time Frame: as for outcome 2
Population: All participants with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
score on a scale
  Post-intervention: number analyzed (Participants) | 54 | 51
  Post-intervention | 44.44 (42.95) | 52.94 (44.81)
  3 Month: number analyzed (Participants) | 42 | 40
  3 Month | 49.21 (41.8) | 61.67 (43.72)
  6 Month: number analyzed (Participants) | 32 | 33
  6 Month | 48.96 (43.16) | 57.58 (40.2)
  9 month: number analyzed (Participants) | 33 | 33
  9 month | 49.49 (44.19) | 52.53 (38.22)
  12 Month: number analyzed (Participants) | 26 | 29
  12 Month | 51.28 (41.34) | 44.83 (41.09)
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-emotional functioning scores from baseline to post-intervention for all study participants; Test type: Superiority; p = 0.0129, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 366; Median Difference (Net) = 12.52, 95% CI 2-sided [2.67 to 22.37], Standard Error of Mean 5.01; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-emotional functioning scores from baseline to 3-month for all study participants; Test type: Superiority; p = 0.0008, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 366; Mean Difference (Net) = 19.84, 95% CI 2-sided [8.32 to 31.36], Standard Error of Mean 5.86; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-emotional functioning scores from baseline to 6-month for all study participants; Test type: Superiority; p = 0.0036, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 366; Median Difference (Net) = 17.99, 95% CI 2-sided [5.92 to 30.06], Standard Error of Mean 6.14; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-emotional functioning scores from baseline to 9-month for all study participants; Test type: Superiority; p = 0.007, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 366; Median Difference (Net) = 16.24, 95% CI 2-sided [4.47 to 28.01], Standard Error of Mean 5.98; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean SF36-emotional functioning scores from baseline to 12-month for all study participants; Test type: Superiority; p = 0.065, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 366; Mean Difference (Net) = 12.26, 95% CI 2-sided [-0.68 to 25.19], Standard Error of Mean 6.58; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: PEERS vs Social Interaction; Null hypothesis: There is no difference in the change of emotional functioning over time between the control and PEERS participants; Test type: Superiority; p = 0.8810, Mixed Models Analysis

5. Secondary Outcome: Cornell Health Service Index - ER Service Use
Description: Health service use is measured with the Cornell Service Index, a questionnaire that includes both clinical and informal community-based health services and has been used in depression care studies among older adults. The index asks whether an individual has used a list of services in the 4 months prior, what type of provider was seen, the site of the service, and reasons for service use. Numbers reported indicate the number of participants who reported hospital and emergency service use at specified timepoints.
Time Frame: as for outcome 1
Population: All participants with at least one assessment completed
Measure: Count of Participants; unit: Participants
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
Participants
  Post-intervention: number analyzed (Participants) | 54 | 51
  Post-intervention | 5 | 8
  3 Month: number analyzed (Participants) | 43 | 42
  3 Month | 12 | 2
  6 Month: number analyzed (Participants) | 33 | 36
  6 Month | 7 | 7
  9 Month: number analyzed (Participants) | 32 | 34
  9 Month | 13 | 9
  12 Month: number analyzed (Participants) | 28 | 29
  12 Month | 4 | 9
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the change in probability of ER use from baseline to post-intervention between PEERS and control participants; Test type: Superiority; p = 0.031, F-test for overall significance — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 370; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Engagement - Adherence
Description: Engagement (adherence) was measured by percentage of attendance of meetings as reported by the peer mentors, with a threshold of 80% of meetings attended.
Time Frame: Intervention 1-8 weeks
Population: All participants with at least one assessment completed
Measure: Count of Participants; unit: Participants
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
Participants
  Week 1: number analyzed (Participants) | 67 | 62
  Week 1 | 67 | 62
  Week 2: number analyzed (Participants) | 64 | 61
  Week 2 | 64 | 61
  Week 3: number analyzed (Participants) | 61 | 60
  Week 3 | 61 | 60
  Week 4: number analyzed (Participants) | 69 | 59
  Week 4 | 61 | 59
  Week 5: number analyzed (Participants) | 60 | 58
  Week 5 | 60 | 58
  Week 6: number analyzed (Participants) | 59 | 56
  Week 6 | 59 | 56
  Week 7: number analyzed (Participants) | 57 | 56
  Week 7 | 57 | 56
  Week 8: number analyzed (Participants) | 57 | 56
  Week 8 | 57 | 56

7. Secondary Outcome: Working Alliance Inventory - Goal
Description: Working alliance was measured on a weekly basis only in the intervention arm with the Working Alliance Inventory-SF. The survey has 12 items with subscales that measure affective bond, and agreement on tasks and goals and are scored using a Likert scale. The goal subscore was calculated by summing items 1, 6, 8, and 11. The subscale ranges from scores of 4-28, with higher scores indicating better agreement on goals.
Time Frame: Intervention weeks 1-8
Population: All participants in the PEERS intervention with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS
Number analyzed (Participants) | 69
score on a scale
  Week 1: number analyzed (Participants) | 39
  Week 1 | 21.85 (5.28)
  Week 2: number analyzed (Participants) | 37
  Week 2 | 23.17 (3.83)
  Week 3: number analyzed (Participants) | 41
  Week 3 | 23.98 (3.81)
  Week 4: number analyzed (Participants) | 41
  Week 4 | 25.05 (2.95)
  Week 5: number analyzed (Participants) | 40
  Week 5 | 24.85 (3.23)
  Week 6: number analyzed (Participants) | 42
  Week 6 | 25.1 (3.22)
  Week 7: number analyzed (Participants) | 43
  Week 7 | 25.63 (3)
  Week 8: number analyzed (Participants) | 41
  Week 8 | 26.21 (2.33)

8. Secondary Outcome: Working Alliance Inventory - Bond
Description: Working alliance was measured on a weekly basis only in the intervention arm with the Working Alliance Inventory-SF. The survey has 12 items with subscales that measure affective bond, and agreement on tasks and goals and are scored using a Likert scale. The bond subscore was calculated by summing items 3, 5, 7, and 9. The subscale ranges from 4-28. A higher subscore indicates higher affective bond.
Time Frame: Intervention weeks 1-8
Population: All participants in the PEERS intervention with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS
Number analyzed (Participants) | 69
score on a scale
  Week 1: number analyzed (Participants) | 39
  Week 1 | 23.28 (5.14)
  Week 2: number analyzed (Participants) | 37
  Week 2 | 24.49 (3.38)
  Week 3: number analyzed (Participants) | 41
  Week 3 | 24.63 (3.31)
  Week 4: number analyzed (Participants) | 41
  Week 4 | 25.02 (2.95)
  Week 5: number analyzed (Participants) | 40
  Week 5 | 25.02 (3.38)
  Week 6: number analyzed (Participants) | 42
  Week 6 | 25.45 (3.02)
  Week 7: number analyzed (Participants) | 43
  Week 7 | 25.51 (2.86)
  Week 8: number analyzed (Participants) | 41
  Week 8 | 26.17 (2.53)

9. Secondary Outcome: Working Alliance Inventory - Task
Description: Working alliance was measured on a weekly basis only in the intervention arm with the Working Alliance Inventory-SF. The survey has 12 items with subscales that measure affective bond, and agreement on tasks and goals and are scored using a Likert scale. The task subscore was calculated by summing items 2, 4, 10, and 12. The subscale ranges from 4-28. A higher subscore indicates higher agreement on tasks.
Time Frame: Intervention weeks 1-8
Population: All participants in the PEERS intervention with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS
Number analyzed (Participants) | 69
score on a scale
  Week 1: number analyzed (Participants) | 38
  Week 1 | 21.24 (4.39)
  Week 2: number analyzed (Participants) | 35
  Week 2 | 20.97 (4.15)
  Week 3: number analyzed (Participants) | 43
  Week 3 | 22.67 (4.12)
  Week 4: number analyzed (Participants) | 38
  Week 4 | 23.13 (4.32)
  Week 5: number analyzed (Participants) | 37
  Week 5 | 23.03 (4.25)
  Week 6: number analyzed (Participants) | 39
  Week 6 | 23.31 (4.11)
  Week 7: number analyzed (Participants) | 41
  Week 7 | 24.12 (3.82)
  Week 8: number analyzed (Participants) | 36
  Week 8 | 24.69 (3.62)

10. Secondary Outcome: UCLA Loneliness Scale
Description: The 20-item R-UCLA loneliness scale measures one's subjective feelings of loneliness as well as feelings of social isolation. Items are summed to create a score. The scores range from 20-80 and higher scores indicating higher level of loneliness. A total score of 20-34 represents low degree of loneliness; 35-49 represent moderate degree of loneliness; 50-64 represent moderately high degree of loneliness; and 65 or above represent high degree of loneliness.
Time Frame: as for outcome 1
Population: All participants with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
score on a scale
  Baseline | 51.54 (15.75) | 47.67 (15.43)
  Post-intervention: number analyzed (Participants) | 54 | 50
  Post-intervention | 44.56 (14.91) | 42.72 (12.69)
  3 Months: number analyzed (Participants) | 42 | 41
  3 Months | 43.9 (13.5) | 39.24 (12.91)
  6 Months: number analyzed (Participants) | 33 | 33
  6 Months | 41.79 (16.24) | 42.52 (13.44)
  9 Months: number analyzed (Participants) | 35 | 34
  9 Months | 43.71 (17.05) | 39.94 (14.12)
  12 Months: number analyzed (Participants) | 29 | 29
  12 Months | 42.93 (17.76) | 40.17 (14.56)
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean UCLA Loneliness scores from baseline to post-intervention for all study participants; Test type: Superiority; p = 0.0005, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 414; Mean Difference (Net) = -4.98, 95% CI 2-sided [-7.78 to -2.18], Standard Error of Mean 1.42 — Score difference: post-intervention - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean UCLA Loneliness scores from baseline to 3-month for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 414; Mean Difference (Net) = -7.38, 95% CI 2-sided [-11.08 to -3.69], Standard Error of Mean 1.88 — Score difference: 3-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean UCLA Loneliness scores from baseline to 6-month for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 414; Mean Difference (Net) = -7.63, 95% CI 2-sided [-11.3 to -3.95], Standard Error of Mean 1.87 — Score difference: 6-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean UCLA Loneliness scores from baseline to 9-month for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 414; Mean Difference (Net) = -8.12, 95% CI 2-sided [-11.53 to -4.7], Standard Error of Mean 1.74 — Score difference: 9-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean UCLA Loneliness scores from baseline to 12-month for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 414; Mean Difference (Net) = -8.26, 95% CI 2-sided [-12.37 to -4.14], Standard Error of Mean 2.09 — Score difference: 12-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no statistical difference in the change of UCLA Loneliness score over time between control and PEERS participants; Test type: Superiority; p = 0.6857, Mixed Models Analysis

11. Secondary Outcome: General Self-Efficacy Scale
Description: The General Self-Efficacy Scale assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. GSES score is calculated by summing all item scores. The score ranges from 10-40 and higher scores indicating more self-efficacy.
Time Frame: as for outcome 1
Population: All participants with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
score on a scale
  Post-intervention: number analyzed (Participants) | 54 | 51
  Post-intervention | 27.98 (5.33) | 27.92 (4.59)
  3 Months: number analyzed (Participants) | 43 | 42
  3 Months | 27.93 (5.21) | 26.62 (3.91)
  6 Months: number analyzed (Participants) | 33 | 35
  6 Months | 26.15 (5.33) | 27.91 (4.06)
  9 Months: number analyzed (Participants) | 36 | 34
  9 Months | 27.39 (4.7) | 28.65 (4.28)
  12 Months: number analyzed (Participants) | 29 | 29
  12 Months | 27.93 (3.8) | 28 (4.93)
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean GSES scores from baseline to post-intervention for all study participants; Test type: Superiority; p = 0.001, Mixed Models Analysis; Degrees of freedom: 421; Mean Difference (Net) = 1.79, 95% CI 2-sided [0.72 to 2.86], Standard Error of Mean 0.54 — Score difference: post-intervention - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean GSES scores from baseline to 3-month for all study participants; Test type: Superiority; p = 0.18, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 421; Mean Difference (Net) = 0.93, 95% CI 2-sided [-0.39 to 2.25], Standard Error of Mean 0.67 — Score difference: 3-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean GSES scores from baseline to 6-month for all study participants; Test type: Superiority; p = 0.11, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 421; Mean Difference (Net) = 1.11, 95% CI 2-sided [-0.24 to 2.45], Standard Error of Mean 0.68 — Score difference: 6-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean GSES scores from baseline to 9-month for all study participants; Test type: Superiority; p = 0.0006, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 421; Mean Difference (Net) = 2.26, 95% CI 2-sided [0.98 to 3.54], Standard Error of Mean 0.65 — Score difference: 9-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean GSES scores from baseline to 12-month for all study participants; Test type: Superiority; p = 0.001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 421; Mean Difference (Net) = 2.48, 95% CI 2-sided [1.01 to 3.95], Standard Error of Mean 0.75 — Score difference: 12-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: PEERS vs Social Interaction; Null hypothesis: There is no difference in the change of GSES scores over time between the control and PEERS participants; Test type: Superiority; p = 0.1195, Mixed Models Analysis

12. Secondary Outcome: Brief COPE - Adaptive Coping
Description: The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. Reliance on adaptive coping strategies were calculated as the sum of the following subscales: active coping (item 2, 7), emotional support (item 5, 15), use of informational support (item 10, 23), positive reframing (item 12, 17), planning (item 14,25), acceptance (item 20, 24), religion (item 22, 27). Each of the subscales ranges from 2-8. The range of scores for adaptive coping is 14-56, with higher scores indicating higher adaptive coping.
Time Frame: as for outcome 1
Population: All participants with at least one assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEERS | Social Interaction
Number analyzed (Participants) | 69 | 65
score on a scale
  Post-intervention: number analyzed (Participants) | 52 | 51
  Post-intervention | 44.12 (8.5) | 41.31 (7.43)
  3 Months: number analyzed (Participants) | 42 | 40
  3 Months | 44.5 (7.86) | 39.62 (7.87)
  6 Months: number analyzed (Participants) | 33 | 32
  6 Months | 42.7 (7.44) | 41.22 (6.99)
  9 Months: number analyzed (Participants) | 33 | 33
  9 Months | 44.36 (8.13) | 42.64 (7.24)
  12 Months: number analyzed (Participants) | 24 | 28
  12 Months | 44.08 (7.78) | 39.57 (9.22)
Statistical Analysis 1: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Brief-COPE Adaptive Coping scores from baseline to post-intervention for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 361; Mean Difference (Net) = 3.22, 95% CI 2-sided [1.71 to 4.73], Standard Error of Mean 0.77 — Score difference: post-intervention - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Brief-COPE Adaptive Coping scores from baseline to 3-month for all study participants; Test type: Superiority; p = 0.0123, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 361; Mean Difference (Net) = 2.59, 95% CI 2-sided [0.57 to 4.62], Standard Error of Mean 1.03 — Score difference: 3-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Brief-COPE Adaptive Coping scores from baseline to 6-month for all study participants; Test type: Superiority; p = 0.01, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 361; Mean Difference (Net) = 2.63, 95% CI 2-sided [0.63 to 4.63], Standard Error of Mean 1.02 — Score difference: 6-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Brief-COPE Adaptive Coping scores from baseline to 9-month for all study participants; Test type: Superiority; p < 0.0001, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 361; Mean Difference (Net) = 4.18, 95% CI 2-sided [2.32 to 6.04], Standard Error of Mean 0.95 — Score difference: 9-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no difference in the mean Brief-COPE Adaptive Coping scores from baseline to 12-month for all study participants; Test type: Superiority; p = 0.0078, Mixed Models Analysis — The a priori threshold for statistical significance is p=0.05; Degrees of freedom: 361; Mean Difference (Net) = 3.14, 95% CI 2-sided [0.83 to 5.44], Standard Error of Mean 1.17 — Score difference: 12-month - baseline; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: PEERS vs Social Interaction; Null hypothesis: there is no statistical difference in the change in adaptive coping over time between control and PEERS participants; Test type: Superiority; p = 0.1408, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data is collected through study completion, an average of 18 months.
Arm/Group | PEERS | Social Interaction
All-Cause Mortality (participants affected / at risk) | 1/75 | 2/74
Serious Adverse Events (participants affected / at risk) | 1/75 | 4/74
Other Adverse Events (participants affected / at risk) | 0/75 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEERS (N=75) | Social Interaction (N=74)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Admission to Hospice (General disorders) | 0 (0) | 1 (1)
Death (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Drop outs leading to small number of subjects analyzed at 12 month follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT04319094/Prot_SAP_000.pdf